CLINICAL TRIAL: NCT00915512
Title: An Open-label, Single-arm, Multicenter, Phase IV Study to Evaluate the Response to Treatment and Safety of Flexible Dose Treatment With Extended-release Paliperidone in Patients With Schizophrenia
Brief Title: A Phase 4 Study to Evaluate Response to Treatment and Safety of Paliperidone Extended-Release in Participants With Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen-Cilag Turkey (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR016543; R076477SCH4027
Record Dates: First submitted 2009-06-05; First posted 2009-06-08 (Estimated); Last update posted 2013-10-10 (Estimated); Status verified 2013-10

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Paliperidone; Invega
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paliperidone extended-release (ER) (Experimental)
  Interventions: Drug: Paliperidone extended-release (ER)

INTERVENTIONS:
Drug: Paliperidone extended-release (ER) — Paliperidone ER tablets will be administered orally once daily as flexible dose ranging from 3 to 12 milligram (mg) per day for 12 months. The recommended dose will be 6 mg once daily.
  Other Names: Invega

SUMMARY:
The purpose of this study is to evaluate the response to treatment and safety of paliperidone extended-release (mechanism to dissolve a drug over time in order to be released slower and steadier into the blood stream) in participants with schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions and hallucinations, and withdrawal into the self).

DETAILED DESCRIPTION:
This is a non-randomized, single-arm, multi-center (conducted in more than one center) study to explore response to treatment and safety of flexible dose of paliperidone extended-release (ER) in participants with schizophrenia. During the study period, dose of paliperidone ER will remain within the range of 3 to 12 milligram per day and will be administered for 12 months. Both hospitalized and non-hospitalized participants may be included in the study. Participants may switch to any effective dose of paliperidone ER from any oral antipsychotic medication without dose adjustment or if required, cross-dose adjustment may be done. Maximum 4 weeks of switching period is allowed. Use of anticholinergic (opposing the actions of the acetylcholine, a neurotransmitter) drugs will not be restricted. Response to treatment will be evaluated primarily through total Personal and Social Performance (PSP) Scale. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia diagnosis according to Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV)
* Recent onset (less than 3 years after the first episode/hospitalization) schizophrenia but either not on antipsychotic medication for at least 3 months or in need of antipsychotic medication switches because of safety and/or lack of efficacy reasons
* To be considered physically healthy at Screening according to vital signs and physical examination findings. If there are abnormalities, they must be consistent with the underlying illness in the study population
* Women at postmenopausal state for at least 1 year; or undergone surgical sterilization, or for women with child-bearing status, should be willing to use an effective contraceptive method throughout the study
* Participants who are willing and capable to complete the questionnaires

Exclusion Criteria:

* Use of clozapine, depot neuroleptics or risperidone within the last 3 months
* Any unstable clinical condition including clinically important abnormal laboratory findings
* Previous and current tardive dyskinesia (abnormal involuntary movements which primarily affect the extremities, trunk, or jaw) symptoms
* History of malignant neuroleptic syndrome
* To be considered carrying high risk regarding adverse effects, homicide and/or suicide

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2009-05; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Total Personal and Social Performance (PSP) Score at Month 12 | Baseline and Month 12
  The PSP is a clinician-rated scale that reflects social functioning in 4 domains of behavior (socially useful activities including work and study, personal and social relationships, self care, and disturbing and aggressive behaviors). The total score ranges from 1 to 100 (score of 71 to 100 will have a mild degree of difficulty; from 31 to 70, varying degrees of disability; less than or equal to 30, functioning so poorly as to require intensive supervision) divided into 10 equal intervals to rate the degree of difficulty (i=absent to vi=very severe) in each of the 4 domains.

SECONDARY OUTCOMES:
Change from Baseline in Global Assessment of Functioning (GAF) Score at Month 12 | Baseline and Month 12
  The GAF is a 100-point tool to measure overall psychological, social and occupational functioning of adults. The higher score range (that is, 91 to 100) refers to a superior functioning in a wide range of activities, and absence of symptoms. The lower score range (that is, 1 to 10) refers to persistent danger of severely hurting self or others; or persistent inability to maintain minimum personal hygiene; or serious suicidal act with clear expectation of death.
Change from Baseline in Total Positive and Negative Syndrome Scale (PANSS) Score and Subscales Score at Month 12 | Baseline and Month 12
  The PANSS is a scale which measures the severity of psychotic symptoms of schizophrenia. Score ranges from 30 to 210 where 30=best and 210=worst. The scale consists of three subscales: positive subscale (Range 7 to 49), negative subscale (Range 7 to 49) and general psychopathology subscale (Range 16 to 112), which measures from absent to extreme condition. Higher scores indicate worsening.
Change from Baseline in Short Form (SF)-36 Scale Score at Month 12 | Baseline and Month 12
  The SF-36 is a survey that measures 8 domains of health including: physical functioning, role limitations due to physical health (role-physical), bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems (role-emotional) and general mental health. Each item is scored on a range of 0 to 100. Worst value is 0 and best value is 100.
Change from Baseline in Percentage of Participants With Relapse at Month 12 | Baseline and Month 12
  The relapse will be diagnosed if participants meet any of the following criteria on 2 consecutive evaluations conducted 3 to 5 days apart: Psychiatric hospitalization; increase in level of care necessary and 25 percent increase in total PANSS score from Baseline; significant clinical deterioration defined as a clinical global impression of change scale score of 6 (indicating much worse); deliberate self-injury; clinically significant suicidal or homicidal ideation; violent behavior resulting in significant injury to another person or property; exceeding the registered dose of drug.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Turkey Clinical Trial, Study Director — Janssen-Cilag Turkey
Locations (7):
- Turkey (Türkiye) (7):
  - Adana
  - Ankara
  - Antalya
  - Bursa
  - Istanbul
  - Manisa
  - Samsun

REFERENCES:
- See also: An open-label, single-arm, multicenter, phase IV study to evaluate the response to treatment and safety of flexible dose treatment with extended-release paliperidone in patients with schizophrenia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=2361&filename=CR016543_CSR.pdf